CLINICAL TRIAL: NCT02994251
Title: A Phase II Trial of Systemic Chemotherapy (Gemcitabine and Cisplatin) in Combination With Conventional Transarterial Chemoembolization (cTACE) in Patients With Advanced Intra-Hepatic Cholangiocarcinoma (ICC)
Brief Title: A Trial of Systemic Chemotherapy in Combination With Conventional Transarterial Chemoembolization in Patients With Advanced Intra-Hepatic Cholangiocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to low enrollment making it unlikely to meet recruitment goals.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1603017367
Record Dates: First submitted 2016-12-06; First posted 2016-12-15 (Estimated); Results first posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Unresectable Intrahepatic Cholangiocarcinoma
MeSH Terms: interventions — Gemcitabine; Cisplatin; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- All subjects (Experimental): Patients must have advanced, unresectable intrahepatic cholangiocarcinoma (ICC) defined as biopsy-confirmed adenocarcinoma in the liver, with an immunohistochemical profile consistent with a pancreatico-biliary primary, not involving the common bile duct or bifurcation, and not amenable to surgical resection.
  Interventions: Drug: gemcitabine; Drug: Cisplatin; Drug: Conventional TACE (transarterial chemoembolization) with Doxorubicin/Mitomycin-C

INTERVENTIONS:
Drug: gemcitabine — 1000 mg/m^2 of gemcitabine on Day 1 and 8, Dosages may be modified or delayed due to toxicities
Drug: Cisplatin — 25 mg/m^2 on Day 1 and 8, Dosages may be modified or delayed due to toxicities
Drug: Conventional TACE (transarterial chemoembolization) with Doxorubicin/Mitomycin-C — If conventional transarterial chemoembolization (TACE) is warranted based on MRI assessment and the patient meets all the eligibility criteria for TACE therapy, then cTACE will be scheduled to take place during Week 3 of that cycle. Patients will always receive the first cTACE for study; follow-up cTACE will occur on demand.

SUMMARY:
The study will be a single-center, single-arm, Phase II study of gemcitabine and cisplatin in combination with conventional trans-arterial chemoembolization therapy in adult patients with advanced ICC. 25 patients will be enrolled over the course of 2 years, with an additional 1.5 years for patient follow-up.

DETAILED DESCRIPTION:
Eligible patients enrolled on study will receive a chemotherapy regimen of gemcitabine and cisplatin administered intravenously on Days 1 and 8 of a 21-day cycle. After every 2 cycles of systemic chemotherapy, patients will receive contrast-enhanced MRI to assess liver disease; conventional trans-arterial chemoembolization (TACE) will be performed as indicated based on this assessment. Patients will receive a maximum of 8 cycles of the gemcitabine/cisplatin combination. Up to 3 TACE treatments may be delivered in this same time frame, with the first TACE taking place after 2 cycles of systemic chemotherapy. Following the treatment period, patients will continue clinical follow-up at 3 month intervals until study exit at 18 months post the start of treatment.

It is hypothesized that the addition of conventional transarterial chemoembolization to standard chemotherapy will result in an improvement in PFS in patients with advanced, unresectable ICC, including patients with extra-hepatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age.
* Patient has advanced, unresectable intrahepatic cholangiocarcinoma (ICC). Advanced, unresectable ICC is defined as biopsy-confirmed adenocarcinoma in the liver, with an immunohistochemical profile consistent with a pancreatico-biliary primary, not involving the common bile duct or bifurcation, and not amenable to surgical resection.
* Eligible for conventional TACE as defined by local treatment guidelines.
* Child-Pugh class of A to B7.
* Adequate end-organ and bone marrow function as manifested as:

  * Hemoglobin ≥ 9 g/dL
  * Absolute neutrophil count ≥ 1500/mm3
  * Creatinine ≤ 2.0 g/dL
  * AST and ALT ≤ 5 x ULN
  * Albumin ≥ 2.4 mg/dL
  * Total bilirubin ≤ 2.5 mg/dL
  * Platelets ≥ 100,000/mm3
  * For TACE procedures, subjects are allowed to have platelets ≥ 75,000/mm3.
* Disease is liver-dominant with >70% of measurable disease burden within the hepatic parenchyma.
* No prior surgery or chemotherapy for ICC.
* ECOG performance status of 0-1.
* No other active malignancy within 2 years.
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of the study.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior or concurrent chemotherapy treatment for advanced ICC.
* History of allergic reactions attributed to compounds of similar chemical or biological composition to gemcitabine, cisplatin, doxorubicin, or mitomycin-C.
* Active treatment with CYP3A4 strong inhibitors or inducers.
* Recent surgical procedure within 21 days of study enrollment.
* Severe and/or uncontrolled co-morbid medical conditions including, but not limited to, active infection, viral hepatitis, congestive heart failure, cardiac arrhythmia, unstable angina pectoris, and psychiatric illness or social circumstance that would limit compliance with study requirements.
* Pregnancy during study duration.
* Active immunosuppressive medications.
* Presence of grade 2 or higher hepatic encephalopathy.
* Complete occlusion of the entire portal venous system. Partial or branch portal vein occlusion allowed if without reversal of flow.
* Radiotherapy within 21 days from treatment with study interventions or medications.
* Current, recent (within 4 weeks of first infusion of this study), or planned participation in additional experimental drug.
* Unstable angina.
* New York Heart Association (NYHA) Grade II or greater congestive heart failure (Appendix C).
* History of myocardial infarction or CVA within 6 months prior to study enrollment.
* Clinically significant peripheral vascular disease.
* Inability to comply with study and/or follow-up procedures.
* Life expectancy of less than 12 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2018-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Schlachter, Principal Investigator — Yale University
Locations (1):
- Smilow Cancer Center, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Subjects
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Confidentiality is a concern as the study was terminated after 1 patient was enrolled, thus any reported data would indicate PHI for this subject.
Arm/Group | All Subjects
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: The primary objective of this study is to evaluate the 12-month progression-free survival (PFS) rate in adult patients with intrahepatic cholangiocarcinoma (ICC) after treatment with gemcitabine and cisplatin in combination with conventional TACE. This is the percentage of patients alive and free of progression at 12-months from enrollment on study. Radiographic assessment of disease burden will be evaluated by mRECIST and qEASL using an MRI scan obtained at the IR clinic visit.
Time Frame: 12 months
Population: Confidentiality is a concern as the study was terminated after 1 patient was enrolled, thus any reported data would indicate PHI for this subject. To prevent this, it was advised to enter 0 as the number of participants analyzed.
Arm/Group | All Subjects
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Survival
Description: Evaluation of overall survival (OS) of adult patients with advanced ICC treated with gemcitabine and cisplatin in combination with conventional TACE. Overall survival is the time from enrollment on study until death of the patient from any cause.
Time Frame: 18 months
Population: as for outcome 1
Arm/Group | All Subjects
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Time to Progression (TTP)
Description: Overall TTP is the time from enrollment on study until radiographic evidence of overall disease progression. Radiographic assessment will be evaluated by mRECIST using MRI every 2 cycles after intra-arterial therapy.
Time Frame: up to 18 months
Population: as for outcome 1
Arm/Group | All Subjects
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Untreatable Progression (TTUP)
Description: TTUP in liver lesions is measured from the time of initiation on cTACE therapy until radiographic evidence of disease progression in targeted lesions. Radiographic assessment will be evaluated by mRECIST using MRI every 2 cycles after intra-arterial therapy.
Time Frame: up to 18 months
Population: as for outcome 1
Arm/Group | All Subjects
Number analyzed (Participants) | 0

5. Secondary Outcome: Toxicities of the Gemcitabine and Cisplatin Regimen in Combination With cTACE Therapy Using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
Description: To evaluate the toxicities of the gemcitabine and cisplatin regimen in combination with cTACE therapy in adult patients with advanced ICC. Safety will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: 18 months
Population: as for outcome 1
Arm/Group | All Subjects
Number analyzed (Participants) | 0

6. Secondary Outcome: Correlation Between Changes in Dynamic Contrast-enhanced MRI of Liver Lesions and Progression Free Survival
Description: early changes in dynamic contrast-enhanced MRI (DCE-MRI) will correlate with long term PFS or OS, specifically as they relate to lesions targeted with cTACE therapy
Time Frame: 18 months
Population: as for outcome 1
Arm/Group | All Subjects
Number analyzed (Participants) | 0

7. Secondary Outcome: Correlation Between Changes in Dynamic Contrast-enhanced MRI of Liver Lesions and Overall Survival
Description: early changes in dynamic contrast-enhanced MRI (DCE-MRI) will correlate with long term OS, specifically as they relate to lesions targeted with cTACE therapy
Time Frame: 18 months
Population: as for outcome 1
Arm/Group | All Subjects
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events collected at baseline until patient exit at 18 months post start of therapy.
Description: Confidentiality is a concern as the study was terminated after 1 patient was enrolled, thus any reported data would indicate PHI for this subject. To prevent this, it was advised to enter 0 as the number of participants analyzed.
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Trial was terminated early due to low enrollment, leading to endpoints not being achievable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT02994251/Prot_SAP_000.pdf